CLINICAL TRIAL: NCT02149407
Title: Efficacy and Safety of Glycerin Suppositories for Treatment of Feeding Intolerance in Very Low Birth Weight Infants
Brief Title: Glycerin Suppositories for Treatment of Feeding Intolerance in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud Medical City (Other Government)
Collaborators: Sulaiman Al Habib Medical Group- Arrayan Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0752
Record Dates: First submitted 2014-05-20; First posted 2014-05-29 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Feeding Intolerance
MeSH Terms: interventions — Glycerol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glycerin group (GG) (Active Comparator): Glycerin group "GG" will receive the 0.5 suppository (700 mg) twice daily for 48 hours. We will use the rounded part and discard the other part then will hold baby's buttocks for 2 minutes to ensure its delivery.
  Interventions: Drug: Glycerin
- Rectal stimulation group (SG) (Active Comparator): Rectal stimulation "SG" by soft cotton swab inserted to around 3 cm. The stick will press against the rectal wall in all direction for 2 minutes twice daily for 48 hours. Ky gel will be used to lubricate the stick and minimize direct friction to rectal wall.
  Interventions: Procedure: Rectal stimulation
- Control group (CG) (Sham Comparator): Control group "CG" will receive routine NICU medical care without any specific intervention for the infant. The research nurse will do shame placebo twice daily by opening his diaper to blind the team for 2 minutes.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Glycerin — Glycerin group "GG" will receive the 0.5 suppository (700 mg) twice daily for 48 hours. We will use the rounded part and discard the other part then will hold baby's buttocks for 2 minutes to ensure its delivery.
  Other Names: Glycerine
  Arms: Glycerin group (GG)
Procedure: Rectal stimulation — Rectal stimulation "SG" by soft cotton swab inserted to around 3 cm. The stick will press against the rectal wall in all direction for 2 minutes twice daily for 48 hours. Ky gel will be used to lubricate the stick and minimize direct friction to rectal wall.
  Arms: Rectal stimulation group (SG)
Other: Control — Control group "CG" will receive routine NICU medical care without any specific intervention for the infant. The research nurse will do shame placebo twice daily by opening his diaper to blind the team for 2 minutes.
  Arms: Control group (CG)

SUMMARY:
Feeding intolerance is a common problem in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with birth weight equal or less than 1500 g

Exclusion Criteria:

* Significant congenital malformations
* Severity of illness such that death is likely in the first few days after birth

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-05 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Time to full feeding (days) | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
  Days to achieve full enteral feeding

SECONDARY OUTCOMES:
Incidence of feeding intolerance | Participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  Feeding intolerance defined as feeding withheld, discontinued, or decreased because the infant was not tolerating enteral feedings.
Incidence of necrotizing enterocolitis (NEC) | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Necrotizing enterocolitis (NEC) defined as per Bell's staging.
Incidence of proven late onset infection | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Incidence of proven late onset infection defined as clinical signs in addition to positive blood culture beyond 72 hours of age.
Incidence of hyperbilirubinemia | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Incidence of hyperbilirubinemia defined as level of bilirubin requiring treatment with phototherapy according to the bilirubin chart used in the participating unit.
Length of hospital stay (days) | At discharge from hospital, an expected average of 8 weeks

OTHER OUTCOMES:
Growth at discharge from hospital | At discharge from hospital, an expected average of 8 weeks
  Growth parameters at discharge from hospital include: Weight (grams), Length (cm), and Head circumference (cm)
Retinopathy of prematurity (ROP) | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Defined by the International Classification of Retinopathy of Prematurity (ICORP)
Bronchopulmonary dysplasia (BPD) | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
Patent ductus arteriosus (PDA) | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  Diagnosed by echocardiogram
Side effects | Participants will be followed for the duration of hospital stay, an expected average of 8 weeks
  For example: Rectal bleeding, Rectal Perforation, or Hematochezia

CONTACTS AND LOCATIONS:
Overall Officials: Latifa Almahmoud, MD, Study Chair — KSMC
Locations (2):
- Saudi Arabia (2):
  - King Saud Medical City, Riyadh
  - Sulaiman Al Habib Medical Group, Riyadh